CLINICAL TRIAL: NCT00553930
Title: Efficacy of Low Dose Pegylated Interferon-α 2a Plus Ribavirin for the Treatment of Chronic Hepatitis C, Genotypes 2 or 3, in HIV-coinfected Patients.
Brief Title: Low Dose Peginterferon-α 2a for Chronic Hepatitis C, Genotypes 2 or 3, in HIV-coinfected Patients
Acronym: SAEI_IFN_1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sociedad Andaluza de Enfermedades Infecciosas (Network)
Responsible Party: Luis F. Lopez-Cortes, Servicio Andaluz de Salud. Hospitales Universitarios Virgen del Rocio
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAEI_IFN_1
Record Dates: First submitted 2007-11-03; First posted 2007-11-06 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Hepatitis C, Chronic; HIV Infections
Keywords: HCV/HIV-coinfected patients; Peginterferon alfa-2a
MeSH Terms: conditions — Hepatitis C, Chronic; HIV Infections | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- G 2/3 (Experimental): Patients with chronic hepatitis or compensated cirrhosis by hepatitis C virus, genotypes 2 or 3, and HIV-coinfected.
  Interventions: Drug: Pegylated interferon alfa-2a and Ribavirin; Drug: Pegylated interferon alfa 2a and Ribavirin

INTERVENTIONS:
Drug: Pegylated interferon alfa-2a and Ribavirin — All patients will be treated with the combination of pegIFN-α 2a (135 μg per week)plus oral Ribavirin at a dose of 800 mg per day. The treatment will be continued up to 20 weeks after reaching an undetectable plasma RNA-HCV. Treatment will be discontinued for patients who did not achieve a reduction of al least 2 log10 IU/ml in plasma HCV RNA levels with respect to baseline at week 12 and will be considered as viral failures.
  Other Names: Pegasys; Copegus
Drug: Pegylated interferon alfa 2a and Ribavirin — Pegylated interferon alfa 2a (135 ug/week)and Ribavirin (800 mg/day). Duration: 20 weeks after reaching an undetectable plasma RNA_HCV. Treatment will be discontinued for patients who did not achieve a decrease of >= 2 log10 IU/ml in plasma HCV RNA levels with respect to baseline at week 12 of treatment or earlier and will be considered as viral failures.
  Other Names: Pegasis (TM); Copegus (TM)

SUMMARY:
Hypothesis: A regimen of low dose of peginterferon alfa-2a plus ribavirin may be as effective as currently recommended regimen for chronic hepatitis C in HIV-coinfected patients.

Objective: To evaluate the efficacy of lower dose of pegylated interferon-α 2a (135 µg weekly) plus ribavirin and a shorter duration of treatment (20 weeks after achieving an undetectable plasmatic HCV-RNA)than the current recommended in patients with chronic hepatitis or compensated cirrhosis by hepatitis C virus, genotypes 2 or 3, in HIV-coinfected patients in real use conditions.

Method: Phase IV, postautorization, open labelled multicenter trial with a planned duration of 118 weeks in which 71 patients from several hospitals of the Servicio Andaluz de Salud will be enrolled. The usual clinical and analytical follow up will be performed but additional blood samples will be obtained for determination of interferon and ribavirin plasma levels. The primary end point wall be a sustained virologic response (defined as an undetectable serum HCV-RNA after 24 weeks after the cessation of treatment). Likewise, rapid virological response (at 4 weeks of treatment), early virological response (at 12 weeks), and end of treatment response rates will be evaluated as well as their relationships with the plasma interferon an ribavirin concentrations determined by ELISA and HPLC, respectively. The safety and tolerability of the studied medications will be evaluated by means of clinical adverse events, physical examination and laboratory results.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* HIV infected, diagnosed with chronic hepatitis or compensated cirrhosis by hepatitis C virus (both anti-HCV antibodies and HCV RNA levels detectable in serum) not previously treated.
* Women of child-bearing age: negative pregnancy test
* Ability to understand and sign a written consent form

Exclusion Criteria:

* Previous interferon treatment
* Pregnancy or breastfeeding
* Acute or chronic hepatitis B infection (positivity for hepatitis B surface antigen or plasma DNA)
* Creatinine clearance < 50 ml/min, according to Cockcroft-Gault
* Decompensated liver disease
* History of organ transplantation
* Concomitant treatment with immunomodulators or didanosine
* Alcohol abuse or use of other recreational drugs
* History of severe psychiatric conditions
* Autoimmune diseases
* Inability to understand and sign a written consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Sustained viral response(undetectable serum HCV-RNA) | 24 weeks after the cessation of treatment

SECONDARY OUTCOMES:
Relationships between the plasma interferon an ribavirin concentrations and efficacy. The safety and tolerability of the studied medications will be evaluated by means of clinical adverse events, physical examination and laboratory results. | Throughout treatment and 24 weeks after finishing it

CONTACTS AND LOCATIONS:
Overall Officials: Luis F Lopez-Cortes, MD, PhD, Study Director — Infectious Disease Service. Hospitales Universitarios Virgen del Rocio. Sevilla. Spain; Antonio Rivero, MD, PhD, Principal Investigator — Hospital Universitario Reina Sofía. Córdoba. Spain; Mercedes Gonzalez, MD, PhD, Principal Investigator — Hospital Universitario Virgen de la Victoria. Malaga. Spain; Angel Garcia, MD, Principal Investigator — Hospital Universitario de Valme. Sevilla. Spain
Locations (1):
- Infectious Diseases Service.Hospitales Universitarios Virgen del Rocio, Seville, Sevilla, Spain

REFERENCES:
- [Derived] Lopez-Cortes LF, Ruiz-Valderas R, Jimenez-Jimenez L, Gonzalez-Escribano MF, Torres-Cornejo A, Mata R, Rivero A, Pineda JA, Marquez-Solero M, Viciana P; Grupo para el Estudio de las Hepatitis Viricas (HEPAVIR) de la Sociedad Andaluza de Enfermedades Infecciosas. Influence of IL28B polymorphisms on response to a lower-than-standard dose peg-IFN-alpha 2a for genotype 3 chronic hepatitis C in HIV-coinfected patients. PLoS One. 2012;7(1):e28115. doi: 10.1371/journal.pone.0028115. Epub 2012 Jan 3. PMID 22235243